CLINICAL TRIAL: NCT04995965
Title: Infections With Enterobacteria Producing Carbapenemases at the University Hospitals of Strasbourg - Descriptive Epidemiology and Risk Factors for Infection in the Event of Colonization
Brief Title: Infections With Enterobacteria Producing Carbapenemases at the University Hospitals of Strasbourg
Acronym: CARBA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8297
Record Dates: First submitted 2021-08-06; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Nfections, Enterobacterial
Keywords: nfections, Enterobacterial; carbapenemases; producers of a carbapenemase

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infections with enterobacteria producing carbapenemases at the University Hospitals of Strasbourg - descriptive epidemiology and risk factors for infection in the event of colonization

There is a worrying situation of an increase in the number of patients colonized with carbapenemase-producing Enterobacteriaceae (CPE) at HUS.

7 to 15% of patients colonized with EPC would develop an infection with EPC. The cohorts published mainly concern patients hospitalized in intensive care. The associated mortality reported in the literature is high (> 25%) and greater than that associated with infection with the same bacterium sensitive to carbapenems.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Subject hospitalized at HUS between 01/01/2011 and 07/31/2021
* Clinical sample or rectal screening smear finding an enterobacterium producing a carbapenemase (EPC)
* Subject not having expressed their opposition to participating in the study

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Subject under guardianship or guardianship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject with clinical sample or rectal screening smear finding an enterobacterium producing a carbapenemase
Sampling Method: Non-Probability Sample
Enrollment: 274 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-01-06 (Estimated); Study Completion 2022-01-06 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of Enterobacteriaceae infections producing carbapenemases | Files analysed retrospectively from January 01, 2011 to July 31, 2021 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Yves HANSMANN, MD, PhD, Principal Investigator — Service de maladies infectieuses et tropicales - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de maladies infectieuses et tropicales - Hôpitaux Universitaires de Strasbourg, Strasbourg, France